CLINICAL TRIAL: NCT03633110
Title: A Phase 1/2a Study to Evaluate the Safety, Tolerability, Immunogenicity, and Antitumor Activity of GEN-009 Adjuvanted Vaccine in Adult Patients With Selected Solid Tumors
Brief Title: Safety, Tolerability, Immunogenicity, and Antitumor Activity of GEN-009 Adjuvanted Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genocea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEN-009-101
Record Dates: First submitted 2018-08-06; First posted 2018-08-16 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Cutaneous Melanoma; Non-small Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck; Urothelial Carcinoma; Renal Cell Carcinoma
Keywords: Vaccine; Personalized; Immunotherapy; Solid Tumor; Personal; Skin; Lung; Cancer; Bladder; Kidney; Melanoma; Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Transitional Cell; Carcinoma, Renal Cell; Neoplasms; Carcinoma | interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Participants in Part A have no evidence of disease when they begin receiving GEN-009 Adjuvanted Vaccine, and have completed treatment with curative intent for their disease (eg, surgical resection, neoadjuvant and/or adjuvant chemotherapy, and/or radiation therapy).
  Part A will consist of approximately 9 participants.
  Interventions: Biological: GEN-009 Adjuvanted Vaccine
- Part B (Experimental): Participants in Part B have advanced or metastatic solid tumors, and will receive GEN-009 Adjuvanted Vaccine in combination with PD-1 inhibitor therapy (nivolumab or pembrolizumab).
  Part B will consist of up to 90 participants.
  Interventions: Biological: GEN-009 Adjuvanted Vaccine; Drug: Nivolumab; Drug: Pembrolizumab

INTERVENTIONS:
Biological: GEN-009 Adjuvanted Vaccine — GEN-009 Adjuvanted Vaccine consists of GEN-009 Drug Product mixed with Hiltonol (poly-ICLC, adjuvant) and is administered by subcutaneous injection.
Drug: Nivolumab — Nivolumab is a PD-1 checkpoint inhibitor approved by the FDA to treat the tumor types in this study.
  Other Names: OPDIVO
  Arms: Part B
Drug: Pembrolizumab — Pembrolizumab is a PD-1 checkpoint inhibitor approved by the FDA to treat the tumor types in this study.
  Other Names: KEYTRUDA
  Arms: Part B

SUMMARY:
In this study, Genocea is evaluating an investigational, personalized adjuvanted vaccine, GEN-009, that is being developed for the treatment of patients with solid tumors. A proprietary tool developed by Genocea, called ATLAS™ (Antigen Lead Acquisition System) will be used to identify neoantigens in each patient's tumor that are recognized by their CD4 and/or CD8 T cells. ATLAS-identified neoantigens will then be incorporated into a patient's personalized vaccine in the form of synthetic long peptides (SLPs).

DETAILED DESCRIPTION:
This first-in-human study of GEN-009 will be conducted in two parts in adult patients with cutaneous melanoma, non-small cell lung cancer (NSCLC), squamous cell carcinoma of the head and neck (SCCHN), urothelial carcinoma, or renal cell carcinoma (Part B only). In Part A, the safety and immunogenicity of single-agent GEN-009 will be evaluated in patients with the above-noted tumor types who have completed treatment with curative intent for their disease (eg, surgical resection, neoadjuvant and/or adjuvant chemotherapy, and/or radiation therapy) and have no evidence of disease (NED) at the time of initiating vaccination with GEN-009. In Part B, up to 15 patients in each disease cohort will be enrolled and evaluated for safety, immunogenicity, and preliminary antitumor activity of GEN-009. Patients in Part B will receive GEN-009 at the schedule selected in Part A, in combination with a PD-1 inhibitor therapy (nivolumab or pembrolizumab) at the approved dose and schedule per the United States Package Insert (USPI). In addition, up to 15 patients who enroll in one of the Part B disease-specific cohorts but whose disease progresses during the screening period therapy may be enrolled into a separate relapsed/refractory disease cohort.

ELIGIBILITY:
General Inclusion Criteria:

* Diagnosis of 1 of the following tumor types:

  1. Melanoma (cutaneous).
  2. NSCLC.
  3. SCCHN (oral, oropharyngeal, hypopharyngeal, or laryngeal).
  4. Urothelial carcinoma.
  5. Renal cell carcinoma (Part B only).
* Understand the study, be willing to comply with all study procedures and sign the informed consent
* Adequate tumor tissue available
* ECOG performance status of 0 or 1
* Negative pregnancy test (females of childbearing potential)
* Agree to use of contraception during the study until at least 90 days after final GEN-009 dose
* Adequate hematologic, liver, and kidney function

Part A-specific Inclusion:

* Have completed or will complete treatment for their disease with curative intent
* Have no evidence of disease

Part B-specific Inclusion:

* Receiving or will initiate treatment with nivolumab or pembrolizumab per disease as listed below:

  1. NSCLC: Patients with metastatic non-squamous NSCLC beginning first-line pembrolizumab in combination with pemetrexed and platinum chemotherapy, or metastatic squamous NSCLC beginning first-line pembrolizumab in combination with carboplatin and either paclitaxel or nab-paclitaxel
  2. SCCHN: Patients beginning pembrolizumab with recurrent or metastatic SCCHN with disease progression on or after a platinum-based therapy, or beginning first-line pembrolizumab for recurrent or metastatic SCCHN if tumors express PD-L1 with a Combined Positive Score (CPS) ≥ 1.
  3. Cutaneous Melanoma: Patients with unresectable or metastatic cutaneous melanoma beginning nivolumab monotherapy or nivolumab in combination with ipilimumab.
  4. Urothelial Carcinoma: Patients with locally advanced or metastatic urothelial carcinoma who are beginning pembrolizumab who:

     1. Are not eligible for cisplatin-containing chemotherapy, and tumor is PD-L1 positive with CPS ≥ 10, or are not eligible for any platinum-containing chemotherapy, OR
     2. Have had disease progression during or following platinum-containing chemotherapy, or within 12 months of neoadjuvant or adjuvant treatment with platinum-containing chemotherapy.
  5. Renal Cell Carcinoma:

     1. Patients with advanced RCC who have received prior anti-angiogenic therapy, and are beginning nivolumab monotherapy, OR
     2. Untreated patients with intermediate or poor risk RCC based on the IMDC score who are beginning nivolumab in combination with ipilimumab.
* Disease assessment by CT or MRI
* Have at least 1 lesion that is measureable by RECIST 1.1
* Agree to a tumor biopsy 50 days after first GEN-009 vaccination
* Participants with hypothyroidism must be on thyroid replacement treatment

General Exclusion Criteria:

* Received a live vaccine ≤ 28 days, or a non-live vaccine ≤ 14 days, prior to the first dose of GEN-009
* Acute or chronic skin disorders that would interfere with injection
* Receiving immunosuppressive therapies or systemic corticosteroids. Note: Use of topical corticosteroids or inhaled corticosteroids is acceptable
* Allergy to the vaccine adjuvant Hiltonol (poly-ICLC)
* Active hepatitis B or hepatitis C infection
* HIV Positive
* History of clinically significant cardiac condition
* History of leptomeningeal carcinomatosis
* Had clinically active immune-mediated disease within 5 years
* Received a prior allogeneic stem cell transplant
* Has primary immune deficiency
* Received a prior solid organ transplant
* Has malignant disease, other than the tumor types being treated in this study
* Female patient who is pregnant, breastfeeding, or who plans to become pregnant from the signing of the informed consent until ≥ 90 days from last dose of GEN-009
* Any condition that in the judgment of the PI would make the patient inappropriate for enrollment in the study
* Patient has received cytotoxic chemotherapy within 4 weeks of the first leukapheresis

Part A-specific Exclusion Criteria:

* Has received or requires more than 2 adjuvant or neoadjuvant regimens (other than surgical excisions) given with curative intent prior to first GEN-009 vaccination
* Has not recovered or stabilized from any clinically significant toxicity associated with any prior procedure or anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1.5 years after first GEN-009 vaccination
  Adverse events will be graded according to the NC Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
T-cell responses to GEN-009 adjuvanted vaccine | 1.5 years after first GEN-009 vaccination
  Immunogenicity based on T-cell responses to GEN-009

SECONDARY OUTCOMES:
Antitumor activity of GEN-009 in Part B | 48 weeks after first GEN-009 vaccination
  Evaluation conducted based on RECIST v1.1 (and immune-related RECIST [irRECIST], where appropriate)

OTHER OUTCOMES:
Long-term clinical outcomes of Part A participants | 1.5 years after first GEN-009 vaccination
  Disease recurrence
Additional cellular responses after vaccination with GEN-009 | 1 year after first GEN-009 vaccination
  Cytokine secretion
Phenotype of circulating immune cells after vaccination with GEN-009 | 1 year after first GEN-009 vaccination
  Measured by flow cytometry
Tumor-infiltrating T cells after vaccination with GEN-009 | 1 year after first GEN-009 vaccination
  Will be examined in tumor biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Arthur P. DeCillis, MD, Study Director
Locations (11):
- United States (11):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - John Wayne Cancer Institute - Providence Saint John's Health Center, Santa Monica, California
  - University of Colorado, Anschutz Cancer Pavilion, Aurora, Colorado
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

REFERENCES:
- See also: OPDIVO (nivolumab) United States Prescribing Information — https://rm2.scinet.fda.gov/druglabel/rs/spl/by-id/242058/242058.html